CLINICAL TRIAL: NCT02209129
Title: 3D Digital Breast Tumorsynthesis Versus 2D Digital Mammography in the Clinical Evaluation of Women at High Risk for Breast Cancer
Brief Title: Digital 3D Breast Tomosynthesis Versus 2D in Clinical Evaluation of High Risk Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Chantal Van Ongeval, MD, Phd, Prof. dr. Van Ongeval Chantal, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: B322201421047
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer
Keywords: digital breast tomosynthesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women at high risk for breast cancer

SUMMARY:
Patients with a higher breast cancer risk (higher than 17% according to the IBIS calculation) will receive a 2D digital mammography together with a 3D tomosynthesis (so called combo tomo) of both breasts in two views in order to investigate the additional value of tomosynthesis in the diagnosis of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* women
* more than 17% risk for breast cancer (IBIS calculation)
* > 40y old

Exclusion Criteria:

* < 40y old

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with an increased risk for breast cancer > 17% according to the IBIS calculation, and also defined by the Multidisciplinary Breast centre UZ Leuven, Belgium
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Tumor dectection rate | 2 years
  The addititional value of 3D tomosythesis to 2D digital mammography will be evaluated by the cancer detection rate, falls negative and falls positive results.

SECONDARY OUTCOMES:
Falls negative, Falls positive results, accuracy | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Van Ongeval, MD,Phd, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium